CLINICAL TRIAL: NCT06914167
Title: The Effectiveness of Lavender Aromatherapy Combined With Slow Breathing Exercises in Improving Occupational Burnout and Sleep Disorders Among Nursing Staff
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chen, Yao-Hsiang, Assistant hand nurse, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TSGH-SS_E_114015
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-03

CONDITIONS: Sleep Wake Disorders
Keywords: Sleep Wake Disorders
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Control Group (No Intervention): Participants will maintain their usual lifestyle without any intervention.
- Breathing-Only Group (Placebo Comparator): Participants will perform slow breathing training (6 breaths per minute) for 3 minutes daily before bedtime, without any essential oil inhalation, for 4 weeks.
  Interventions: Behavioral: Slow Breathing Exercises
- Experimental Group 1 (Experimental): Participants will receive slow breathing training (6 breaths per minute) once daily before bedtime, combined with the inhalation of 3 drops of natural lavender essential oil on a towel, for 3 minutes, over a 4-week period.
  Interventions: Behavioral: Slow Breathing Exercises; Behavioral: Lavender Essential Oil Inhalation
- Experimental Group 2 (Experimental): Same breathing protocol as above, with 3 drops of linalyl acetate-containing essential oil on a towel, for 3 minutes, over a 4-week period.
  Interventions: Behavioral: Slow Breathing Exercises; Behavioral: linalyl acetate essential oil Inhalation
- Experimental Group 3 (Experimental): Same breathing protocol, with 3 drops of linalool-containing essential oil on a towel, for 3 minutes, over a 4-week period.
  Interventions: Behavioral: Slow Breathing Exercises; Behavioral: linalool essential oil Inhalation

INTERVENTIONS:
Behavioral: Slow Breathing Exercises — Participants will perform slow breathing (6 breaths/min) for 3 minutes daily before bedtime
  Arms: Breathing-Only Group; Experimental Group 1; Experimental Group 2; Experimental Group 3
Behavioral: Lavender Essential Oil Inhalation — inhalation of 3 drops of lavender essential oil on a towel,
  Arms: Experimental Group 1
Behavioral: linalyl acetate essential oil Inhalation — inhalation of 3 drops of linalyl acetate essential oil on a towel.
  Arms: Experimental Group 2
Behavioral: linalool essential oil Inhalation — inhalation of 3 drops of linalool essential oil on a towel.
  Arms: Experimental Group 3

SUMMARY:
This study investigates the effects of breathing exercises combined with lavender essential oil inhalation on occupational burnout and sleep disturbances in rotating shift nurses.

DETAILED DESCRIPTION:
This study will adopt a randomized controlled trial (RCT) design targeting rotating shift nurses with at least six months of clinical experience at a regional teaching hospital in northern Taiwan. Eligible participants who consent to join the study will be randomly assigned into five groups using block randomization. The randomization process will be conducted via sealed envelopes to allocate participants into the following groups: Experimental Group 1, Experimental Group 2, Experimental Group 3, Breathing-Only Group, and Control Group.

Experimental Group 1: Participants will receive slow breathing training (6 breaths per minute) once daily before bedtime, combined with the inhalation of 3 drops of natural lavender essential oil on a towel, for 3 minutes, over a 4-week period.

Experimental Group 2: Same breathing protocol as above, with 3 drops of linalyl acetate-containing essential oil.

Experimental Group 3: Same breathing protocol, with 3 drops of linalool-containing essential oil.

Breathing-Only Group: Participants will perform slow breathing training (6 breaths per minute) for 3 minutes daily before bedtime, without any essential oil inhalation, for 4 weeks.

Control Group: Participants will maintain their usual lifestyle without any intervention.

The outcomes will be evaluated using a nurse burnout scale and a sleep quality scale. Measurements will be taken at three time points: baseline (pre-test), 4 weeks after the intervention (post-test 1), and 8 weeks after the intervention (follow-up/post-test 2).

The study is co-led by Yao-Hsiang Chen, Assistant Head Nurse at Tri-Service General Hospital Songshan Branch, and Professor Chia-Hui Lin, School of Nursing, National Defense Medical Center.

ELIGIBILITY:
Inclusion Criteria:

Aged between 20 and 65 years Registered nurses with at least 6 months of clinical experience and currently working rotating shifts Scores ≥1 in each of the three dimensions (emotional exhaustion, reduced personal accomplishment, depersonalization) on the Nursing Burnout Scale (NBS) Willing to participate in the study and accept random assignment

Exclusion Criteria:

Nurses with less than 6 months of clinical experience Individuals with anosmia or reduced sense of smell Diagnosed with psychiatric disorders Allergic to lavender essential oil Not currently working rotating shifts

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Nursing Burnout Scale, NBS | At baseline, and at 4 and 8 weeks following the start of intervention
  The Nurse Burnout Inventory is specifically developed based on nurses' clinical practice experiences. It includes items that reflect three key dimensions: emotional exhaustion resulting from the high-tension clinical work environment, reduced personal accomplishment associated with feelings of ineffectiveness in medical care, and depersonalization, characterized by indifference toward others due to prolonged burnout.

SECONDARY OUTCOMES:
The Chinese version of the Pittsburgh Sleep Quality Index, CPSQI | At baseline, and at 4 and 8 weeks following the start of intervention
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-reported questionnaire designed to assess sleep quality over the past month. It evaluates multiple aspects of sleep, including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. A higher score indicates poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Songshan Branch, Taipei City, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bavarsad NH, Bagheri S, Kourosh-Arami M, Komaki A. Aromatherapy for the brain: Lavender's healing effect on epilepsy, depression, anxiety, migraine, and Alzheimer's disease: A review article. Heliyon. 2023 Jul 20;9(8):e18492. doi: 10.1016/j.heliyon.2023.e18492. eCollection 2023 Aug. PMID 37554839
- [Background] Sugawara Y, Shigetho A, Yoneda M, Tuchiya T, Matumura T, Hirano M. Relationship between mood change, odour and its physiological effects in humans while inhaling the fragrances of essential oils as well as linalool and its enantiomers. Molecules. 2013 Mar 13;18(3):3312-38. doi: 10.3390/molecules18033312. PMID 23486108
- [Background] Zangaro GA, Dulko D, Sullivan D, Weatherspoon D, White KM, Hall VP, Squellati R, Donnelli A, James J, Wilson DR. Systematic Review of Burnout in US Nurses. Nurs Clin North Am. 2022 Mar;57(1):1-20. doi: 10.1016/j.cnur.2021.11.001. PMID 35236600
- [Background] Zaccaro A, Piarulli A, Melosini L, Menicucci D, Gemignani A. Neural Correlates of Non-ordinary States of Consciousness in Pranayama Practitioners: The Role of Slow Nasal Breathing. Front Syst Neurosci. 2022 Mar 21;16:803904. doi: 10.3389/fnsys.2022.803904. eCollection 2022. PMID 35387390
- [Background] Yang CP, Yang CC, Tsai IJ, Lin TH, Chiou YL, Wang HF, Chang CM, Yih KH. The immediate effects of lavender-based essential oil inhalation on subsequent polysomnography in people with poor sleep quality. J Chin Med Assoc. 2023 Jul 1;86(7):665-671. doi: 10.1097/JCMA.0000000000000932. Epub 2023 Apr 25. PMID 37098173
- [Background] Sullivan V, Hughes V, Wilson DR. Nursing Burnout and Its Impact on Health. Nurs Clin North Am. 2022 Mar;57(1):153-169. doi: 10.1016/j.cnur.2021.11.011. Epub 2022 Feb 9. PMID 35236605
- [Background] Moghadam ZE, Delmoradi F, Aemmi SZ, Vaghee S, Vashani HB. Effectiveness of aromatherapy with inhaled lavender essential oil and breathing exercises on ECT-related anxiety in depressed patients. Explore (NY). 2022 Nov-Dec;18(6):683-687. doi: 10.1016/j.explore.2021.12.006. Epub 2021 Dec 30. PMID 35027302
- [Background] Laborde S, Allen MS, Borges U, Dosseville F, Hosang TJ, Iskra M, Mosley E, Salvotti C, Spolverato L, Zammit N, Javelle F. Effects of voluntary slow breathing on heart rate and heart rate variability: A systematic review and a meta-analysis. Neurosci Biobehav Rev. 2022 Jul;138:104711. doi: 10.1016/j.neubiorev.2022.104711. Epub 2022 May 24. PMID 35623448
- [Background] Hedigan F, Sheridan H, Sasse A. Benefit of inhalation aromatherapy as a complementary treatment for stress and anxiety in a clinical setting - A systematic review. Complement Ther Clin Pract. 2023 Aug;52:101750. doi: 10.1016/j.ctcp.2023.101750. Epub 2023 Apr 5. PMID 37031643
- [Background] Balban MY, Neri E, Kogon MM, Weed L, Nouriani B, Jo B, Holl G, Zeitzer JM, Spiegel D, Huberman AD. Brief structured respiration practices enhance mood and reduce physiological arousal. Cell Rep Med. 2023 Jan 17;4(1):100895. doi: 10.1016/j.xcrm.2022.100895. Epub 2023 Jan 10. PMID 36630953
- [Background] Antczak-Komoterska A, Haor B, Malinowska M, Grzelak L, Biercewicz M, Kochman D, Krajewska K, Filipska-Blejder K, Wisniewski A, Slusarz R. Analysis of the Level of Stress and Methods of Coping with Stress among the Nursing Staff. Nurs Rep. 2023 Sep 14;13(3):1318-1330. doi: 10.3390/nursrep13030111. PMID 37755354